CLINICAL TRIAL: NCT03567681
Title: An Exploratory Randomized Open Comparison of Oxtellar XR® vs Oxcarbazepine IR (Trileptal®) for the Treatment of Bipolar Depression
Brief Title: Comparison of Two Forms of Oxcarbazepine for the Treatment of Bipolar Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Collaborative Care Initiative, LLC (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI-BD-001
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Bipolar Depression; Treatment Effectiveness; Measure-based Guidance
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Open randomization to parallel treatment groups
Masking Description: Outcome will be assessed by computer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended release oxcarbazepine (Experimental): Six week of open treatment with extended release oxcarbazepine (Oxtellar XR)
  Interventions: Drug: Extended release oxcarbazepine vs Immediate release oxcarbazepine
- Immediate release oxcarbazepine (Experimental): Six week of open treatment with Immediate release oxcarbazepine ( Trileptal)
  Interventions: Drug: Extended release oxcarbazepine vs Immediate release oxcarbazepine

INTERVENTIONS:
Drug: Extended release oxcarbazepine vs Immediate release oxcarbazepine — Extended release oxcarbazepine vs Immediate release oxcarbazepine
  Other Names: Oxtellar vs Trileptal

SUMMARY:
Consenting subjects with Bipolar depression will remain under the care of their local (psychiatric) care provider and be randomized to a six week course of one of two forms of oxcarbazepine (extended release or immediate release. Study outcomes will be assessed based on outcome measures administered to the subject at home by a computer simulated rater. Local care providers will receive "pre-assessment" reports ahead of each clinical visit, rate the Clinical Global Impression for Severity, and evaluate adverse effects. The primary outcome variable is "treatment effectiveness" operationally defined as the response rate X the completion rate.

DETAILED DESCRIPTION:
This study will use the CCI Engaged Practice platform (EngagedPractice.Com) and will be conducted by a central "meta-site" reviewing eligibility, obtaining consent, randomizing subjects to treatment groups, training local care providers (LCP) to function as sub- investigators and monitoring outcomes.

Subjects will be randomized to six weeks of treatment with extended release oxcarbazepine or immediate release oxcarbazepine,while remaining under the care of their existing LCP.

LCP's will receive sub-investigator training for Good Clinical Practice, Human subjects protection, and all protocol specified assessments and procedures.

A computer simulated rater will collect outcomes (including MADRS, YMRS, PHQ-9, and adverse effects) ahead of each routine clinical visit and provide Measure-based Guidance o the LCP in the form of pre-assessment reports. The primary outcome variable is "treatment effectiveness" operationally defined as the response rate X the completion rate.

ELIGIBILITY:
Inclusion Criteria: The protocol is designed to collect evidence from subjects during the course of routine clinical care. Enrollment is limited to consenting subjects with a current local care provider who agrees that oxcarbazepine is a reasonable next step in managing their bipolar depression

1. Adults male or female, 18-65 years of age, inclusive, at the time of informed consent.
2. Able to access the internet for computer administered ratings.
3. Lifetime mood disorder Diagnosis of Bipolar disorder I or II and a current episode meeting criteria for MDE with or without mixed features according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) at screen and baseline and confirmed by the Collaborative Care Initiative (CCI) review of pre-assessment including bipolarity index score ≥ 50,
4. Severity of current MDE at least moderate depression as defined by Montgomery Asberg Depression Rating Scale (MADRS) ≥20 and least three symptoms of DSM 5 MDE criteria meet threshold for counting toward a current MDE diagnosis (item scores ≥4) at screen and baseline.
5. Duration of current MDE at baseline is at least 4 weeks in and no longer than 2 years
6. Cycle frequency does not exceed 8 mood episodes in the past 365 days.
7. Current treatment regimen stable for at least 4 weeks and must include at least one of three acceptable medication types, but no more than 1 from each class: lithium, one dopamine-blocking agent, one standard antidepressant medication.
8. The LCP agrees that treatment with oxcarbazepine is appropriate, completes study training, and agrees to complete all protocol management and record keeping requirements.
9. Any urine toxicology screens for drugs of abuse (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, and cannabinoids) and alcohol in the 6 months prior to the baseline visit have been negative. Note any positive test result(s) for benzodiazepines accompanied by confirmation of a prescription for a valid medical reason will be allowed.
10. Negative urine pregnancy test at screen or baseline visit.
11. Sexually active women, unless surgically sterile (at least six months prior to study drug administration) or at least one year post-menopausal, must have used an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of condom with spermicide by sexual partner or sterile [at least six months prior to study drug administration] sexual partner) for at least four weeks prior to study drug administration, and must have agreed to continue using such precautions through the End of Study visit. Cessation of birth control after this point was to be discussed with a responsible physician.
12. At least one set of clinical labs including serum sodium, creatinine and TSH have been obtained and within normal limits within the 3 months prior to the baseline visit.

Exclusion Criteria:

1. Inability to provide informed consent in English
2. Current or lifetime diagnosis of epilepsy
3. Pregnancy, breastfeeding or refusal to use birth control
4. Another current Axis I diagnosis that is the primary focus of current treatment
5. Substance or alcohol abuse/dependence at least 6 months prior enrollment
6. Clinically significant abnormal results on clinical laboratories (including serum Creatinine, Sodium, and TSH) at baseline visit or within the prior 3 months.
7. Has started treatment with an FDA approved agent for Bipolar depression within the past 4 weeks
8. Has received treatment with a long-acting injectable antipsychotic or electroconvulsive therapy during the 2 months prior screening
9. If psychotropic medication outside of study limits is required (Note: Subjects may receive any concomitant medications prescribed by their local care providers with the following specific exceptions: Anti-anxiety medications (anxiolytics) exceeding equivalent of lorazepam 2 mg/d.
10. Any long-acting injectable antipsychotic, More than one dopamine blocking agent, More than one standard antidepressant agent, FDA approved treatments for Bipolar depression (quetiapine, lurasidone, the combination of olanzapine and fluoxetine), or Electroconvulsive therapy.)
11. Last dose of another anticonvulsant agent taken in the current week or within 5 half-lives of discontinuation (whichever is longer) prior to enrollment in the study
12. Current treatment requires ongoing anti-anxiety medications (Anxiolytics) exceeding equivalent of lorazepam 2 mg/d.
13. Use of oxcarbazepine (OXC) for treatment of current episode
14. Previous known hypersensitivity to OXC or other related drugs, such as carbamazepine.
15. History or presence of clinically significant, chronic medical condition, (e.g., hyponatremia, any neurological, gastrointestinal, endocrine, cardiovascular, pulmonary, hematological, immunologic, renal, hepatic or metabolic disease) that in the opinion of the clinician or investigator may affect the safety of the subject and the participation to the trial.
16. Active Suicidality (MADRS item 10 >4) Active suicidal plan/intent or active suicidal thoughts in the past 6 months. Any suicide attempt within two years of the screening assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-13 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Effectiveness | 6 weeks
  Treatment Effectiveness is defined as Response Rate (Change from Baseline MADRS > or = 50%) X Completion Rate (completes week 6 of protocol while remaining on assigned treatment).

SECONDARY OUTCOMES:
Tolerability | 6 weeks
  Tolerability is defined as the rate of completion without severe adverse effects reported by subject or clinician. The subject will complete an adverse effects self-report module as part of their "Online Pre-assessment" 1-3 days prior to each clinical visit. The clinician will review the pre-assessment and complete their own adverse effect report at each visit. Items rated as severe by either the subject or the clinician will will be counted as severe. Subjects who remain on study medication for 6 weeks without severe adverse effects will be scored as tolerating treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dauten Family Center for Bipolar Treatment Innovation, Boston, Massachusetts, United States

REFERENCES:
- [Background] Benedetti A, Lattanzi L, Pini S, Musetti L, Dell'Osso L, Cassano GB. Oxcarbazepine as add-on treatment in patients with bipolar manic, mixed or depressive episode. J Affect Disord. 2004 Apr;79(1-3):273-7. doi: 10.1016/S0165-0327(02)00407-X. PMID 15023507
- [Background] Ghaemi SN, Berv DA, Klugman J, Rosenquist KJ, Hsu DJ. Oxcarbazepine treatment of bipolar disorder. J Clin Psychiatry. 2003 Aug;64(8):943-5. doi: 10.4088/jcp.v64n0813. PMID 12927010
- [Background] Sachs GS, Nierenberg AA, Calabrese JR, Marangell LB, Wisniewski SR, Gyulai L, Friedman ES, Bowden CL, Fossey MD, Ostacher MJ, Ketter TA, Patel J, Hauser P, Rapport D, Martinez JM, Allen MH, Miklowitz DJ, Otto MW, Dennehy EB, Thase ME. Effectiveness of adjunctive antidepressant treatment for bipolar depression. N Engl J Med. 2007 Apr 26;356(17):1711-22. doi: 10.1056/NEJMoa064135. Epub 2007 Mar 28. PMID 17392295
- [Background] Morris DW, Trivedi MH. Measurement-based care for unipolar depression. Curr Psychiatry Rep. 2011 Dec;13(6):446-58. doi: 10.1007/s11920-011-0237-8. PMID 21935633
- See also: Platform for assessment and Measure-based Guidance — http://EngagedPractice.com